CLINICAL TRIAL: NCT07243301
Title: Comparison of Thread Embedding Acupuncture at the First Lumbar EX-B2 Point With Sham Thread Embedding Acupuncture on Acute Pain and Quality of Life After Laparoscopic Living Donor Nephrectomy
Brief Title: Thread Embedding Acupuncture vs Sham on Acute Pain and Quality of Life After Laparoscopic Nephrectomy of Living Donor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Salman Matoaya Bustan, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 24-12-1864
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain; Kidney Transplant; Complications
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The intervention group will receive thread implantation acupuncture, while the control group will receive sham thread implantation acupuncture.
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding will be applied to participants and outcome assessors. Group allocation will not be disclosed to them to minimize assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Thread implantation acupuncture
  Interventions: Device: Thread implantation acupuncture
- Control Group (Sham Comparator): Sham thread implantation acupuncture
  Interventions: Device: Sham thread implantation acupuncture

INTERVENTIONS:
Device: Thread implantation acupuncture — Thread implantation acupuncture performed bilaterally at EX-B2 (L1) using polydioxanone (PDO) thread (26G × 38 mm) inserted subcutaneously to a depth of approximately 1-1.5 cm. The procedure is conducted once under aseptic conditions before surgery, combined with standard postoperative analgesic therapy.
  Arms: Intervention Group
Device: Sham thread implantation acupuncture — Sham thread embedding acupuncture performed bilaterally at EX-B2 (L1) using a blunt needle without thread insertion, mimicking the procedure but without embedding material. Participants also receive standard postoperative therapy.
  Arms: Control Group

SUMMARY:
This randomized, double-blind controlled study aims to evaluate the effectiveness of thread implantation acupuncture at EX-B2 L1 in reducing postoperative pain and improving quality of life in patients undergoing laparoscopic living donor nephrectomy. Thirty-four participants will be randomly assigned to receive either thread implantation acupuncture with polydioxanone (PDO) thread at EX-B2 L1 plus standard postoperative therapy or sham thread implantation acupuncture without thread insertion plus the same standard therapy. Pain intensity will be assessed using the Visual Analogue Scale (VAS) and quality of life with the Short-Form 36 (SF-36). The study seeks to determine whether thread implantation acupuncture provides additional analgesic and quality-of-life benefits beyond standard postoperative care.

DETAILED DESCRIPTION:
Laparoscopic donor nephrectomy is the preferred technique for kidney donation due to its minimally invasive nature and faster recovery. However, postoperative pain and decreased quality of life remain significant issues. Excessive reliance on pharmacological analgesia can lead to adverse effects such as hepatotoxicity and gastrointestinal symptoms.

Thread implantation acupuncture involves inserting a biodegradable polydioxanone (PDO) thread into acupuncture points to provide prolonged stimulation. The EX-B2 (L1) point has been shown to modulate lumbar innervation and may help reduce nociceptive signaling associated with postoperative pain.

This double-blind randomized controlled trial compares the analgesic and quality-of-life outcomes between patients receiving thread implantation acupuncture at EX-B2 (L1) plus standard therapy and those receiving sham thread implantation acupuncture plus standard therapy. Pain intensity (VAS) will be measured pre-intervention (Day 0), then at postoperative Days 1, 2, 3, and 14. Quality of life (SF-36) will be evaluated at Day 0 and Day 14. The results are expected to strengthen evidence for thread implantation acupuncture as an adjunctive therapy for acute postoperative pain management and recovery after laparoscopic donor nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Living kidney donors scheduled to undergo laparoscopic living donor nephrectomy.
* Aged 21-60 years.
* Willing to participate and able to sign written informed consent

Exclusion Criteria:

* Hypersensitivity to thread-embedding acupuncture (TEA).
* History of keloid formation or tendency to develop keloids.
* Skin disorders at or near the planned TEA insertion sites.
* Neurological abnormalities or lower-limb deficits on physical examination.
* History of spinal surgery or scheduled for spinal surgery within the next 7 months.
* Scoliosis based on clinical examination.
* Other causes of low back pain, such as inflammatory spondylitis, spinal infection, or tumor.
* Planning to become pregnant within 7 months after LNDH.
* Body Mass Index (BMI) < 18 kg/m².
* Uncontrolled diabetes mellitus.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity (Visual Analogue Scale) | From baseline to postoperative Day 14
  Visual Analogue Scale (0-100 mm) measured at Day 0 (baseline), Day 1, 2, 3, and 14 post-surgery.

SECONDARY OUTCOMES:
Change in Quality of Life (Short Form-36) | Baseline and Day 14.
  Short Form-36 questionnaire assessing eight domains of quality of life at Day 0 and Day 14.
Analgesic Use | Day 0-14.
  Total postoperative paracetamol dose used within 14 days.
Adverse Events Adverse Events Adverse Events | Up to Day 14
  Frequency and type of adverse reactions (pain, bruising, infection, thread extrusion).

CONTACTS AND LOCATIONS:
Overall Officials: KEPK FKUI-RSCM, Principal Investigator — The Health Research Ethics Commitee - Faculty of Medicine Universitas Indonesia and Dr. Cipto Mangunkusumo National Hospital
Locations (1):
- Universitas Indonesia, Jakarta Pusat, Dki Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No